CLINICAL TRIAL: NCT01959074
Title: The Effect of Naftopidil for the Double-J Stent Discomfort: Multicenter, Randomized, Double-blind, Placebo Controlled Study
Brief Title: The Effect of Naftopidil for the Double-J Stent Discomfort
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Chang Wook Jeong, M.D, Ph.D., Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SNUH-URO-2012-04; SNUH-URO-2012-04-DJ (Other: SNU Hosptial IRB)
Record Dates: First submitted 2013-09-24; First posted 2013-10-09 (Estimated); Last update posted 2015-12-10 (Estimated); Status verified 2015-12

CONDITIONS: Disorder of Urinary Stent
MeSH Terms: interventions — naftopidil; aceclofenac

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Naftopidil (Active Comparator): This interventional group will receive analgesics and naftopidil 75mg po qd.
  Interventions: Drug: Naftopidil; Drug: Standard treatment
- Control groups with only analgesics (Placebo Comparator): Control groups will receive only analgesics
  Interventions: Drug: Placebo for Naftopidil; Drug: Standard treatment

INTERVENTIONS:
Drug: Naftopidil — Naftopidil 75mg 1T qd hs
  Other Names: Flivas(TM) in South Korea
  Arms: Naftopidil
Drug: Placebo for Naftopidil — Placebo 1T qd hs
  Arms: Control groups with only analgesics
Drug: Standard treatment — aceclofenac 100mg on demand
  Other Names: Aceclofenac

SUMMARY:
This study is To confirm the efficacy of Naftopidil for reducing discomfort of ureteral stent after urinary stone surgery.

DETAILED DESCRIPTION:
1. Enrollment

   1. patients underwent Double-J ureteral stent indwelling after urological surgery during less than 15 days
   2. patients aged more than 20 years
2. Randomization

   1. naftopidil 75 mg qd or placebo until Double-J stent removal
   2. Standard treatment with pain-killers on demand were also applied.(aceclofenac)
3. Follow-up to the day of Double-J stent removal (Evaluation should be done at stent removal)

ELIGIBILITY:
Inclusion Criteria:Patients to be undergone double-J stent indwelling

* >= 20 years
* undergoing unilateral retrograde double J (DJ) stent placement planned for 5-15 days indwelling

Exclusion Criteria:

* after percutaneous nephrolithotomy, open or laparoscopic ureterolithotomy presence of ureteral stone
* renal insufficiency (serum Cr > 1.4)
* febrile urinary tract infection (fever > 38.0°C, evidence of urinary infection )
* pregnancy or breast feeding
* solitary kidney
* hypersensitivity to Naftopidil
* current use of any alpha blocker, calcium channel blocker, corticosteroid moderate or sever cardiovascular or cerebrovascular disease
* hepatic dysfunction
* prior history of pelvic surgery or irradiation
* prior history of transurethral resection of bladder tumor or prostate surgery
* significant active medical illness which in the opinion of the investigator would preclude protocol treatment
* genetic disorder such ad galactose intolerance, lapp lactase deficiency, glucose-galactose malabsorption

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-05; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Ureteral Stent Symptom Questionaire(USSQ) urinary symptom score | at the day of DJ stent removal, an expected average of 10 days (range: 5-15 days)
  DJ stent removal should be done between study day 5 and 15.
USSQ body pain score | at the day of DJ stent removal, an expected average of 10 days (range: 5-15 days)

SECONDARY OUTCOMES:
USSQ general health score | at the day of DJ stent removal, an expected average of 10 days (range: 5-15 days)
USSQ work performance score | at the day of DJ stent removal, an expected average of 10 days (range: 5-15 days)
USSQ sexual matters score | at the day of DJ stent removal, an expected average of 10 days (range: 5-15 days)
International Prostate Symptom Score(IPSS), QoL score | at the day of DJ stent removal, an expected average of 10 days (range: 5-15 days)
Total analgesics use | at the day of DJ stent removal, an expected average of 10 days (range: 5-15 days)

CONTACTS AND LOCATIONS:
Overall Officials: Chang Wook Jeong, M.D., Ph.D., Principal Investigator — Seoul National University Hospital
Locations (6):
- South Korea (6):
  - Seoul National University Bundang Hospital, Seongnam, Kyunggi
  - Kangwon National University Hospital, Chuncheon
  - Donguk University Ilsan Hospital, Goyang
  - Seoul National University Hospital, Seoul
  - National Medical Center, Seoul
  - Seoul National University Boramae Hospital, Seoul